CLINICAL TRIAL: NCT04827186
Title: Spleen Transplant as an Immunomodulatory Strategy in Solid Organ Transplantation
Brief Title: Spleen Transplant in Solid Organ Transplantation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We did not enroll subjects. If we want, we will open this again at a later date.
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Ivo G Tzvetanov, Chief of Transplantation & Associate Professor, Department of Surgery, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0286
Record Dates: First submitted 2021-03-30; First posted 2021-04-01 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Kidney Transplant Rejection; Positive FCXM (T or B Cell Positive); Positive CDC Cross-Match (B Cell Positive); Kidney/Pancreas Transplant Rejection

STUDY DESIGN:
Intervention Model Description: The protocol presented a single center, open label, prospective trial in which subjects, highly sensitized recipients with a positive T and B flow or positive B standard crossmatch, will undergo spleen transplant and kidney or simultaneous kidney pancreas transplant at the University of Illinois at Chicago. The expected number of patients is 40. Graft and patient survival will be monitored and compared with an historical cohort of highly sensitized patient which received kidney or simultaneous kidney pancreas transplant alone without spleen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- highly sensitized patients with either a positive FCXM, or positive CDC cross-match (Experimental): highly sensitized patients that receive a donor offer and have either a positive FCXM (T or B cell positive) or positive CDC cross-match (B cell positive); a positive CDC cross-match (T cell positive) remains a contraindication at this time.
  Interventions: Procedure: Spleen Transplantation/Removal
- historical cohort of highly sensitized patients with a positive FCXM, or positive CDC cross-match (No Intervention): The control group, as comparison, will be an historical cohort of highly sensitized patients with positive flow (B and T) or positive B standard crossmatch, which received kidney transplant alone or simultaneous kidney and pancreas transplant and followed our standard protocol

INTERVENTIONS:
Procedure: Spleen Transplantation/Removal — Spleen transplantation/removal and kidney transplantation alone or simultaneous kidney and pancreas transplantation in highly sensitized patients with either a positive flow cytometry cross-match (FCXM) (T or B cell positive) or a complement-dependent cytotoxicity (CDC) cross-match (B cell positive).
  Arms: highly sensitized patients with either a positive FCXM, or positive CDC cross-match

SUMMARY:
Although the notions that kidney transplantation is the treatment of choice for patients with end-stage renal disease and that simultaneous kidney and pancreas transplant is the only treatment able to restore euglycemia in patients with type 1 diabetes and selected patients with type 2 diabetes, are now consolidated, rates of transplantation remain low among potential candidates with high levels of preformed anti-HLA antibodies. Most of the data comes from the experience in kidney transplant but can be easily translated to pancreas transplant.

Approximately 30% of patients on the transplant waiting list have evidence of sensitization in the form of alloantibodies, generated from exposure to previous transplants, blood transfusions, pregnancy, or other events. The presence of a panel-reactive antibody level of at least 80% (i.e. a high level of sensitization) creates difficulty in finding matched kidneys from compatible donors, leading to lower rates of transplantation in highly sensitized candidates compared to non-sensitized; the longer waiting times translates in an increased mortality rate. Despite the development of desensitization strategies and the advancement in immunosuppression protocols, it is apparent that transplanting these patients carries an increased risk of acute antibody mediated rejection; 25%-50% of transplants will have an early acute antibody mediated rejection . Most of these rejections can be successfully treated, but a high rate of transplant glomerulopathy and chronic antibody mediated rejection (AMR) leading to accelerated allograft failure is common.

DETAILED DESCRIPTION:
Although the notions that kidney transplantation is the treatment of choice for patients with end-stage renal disease and that simultaneous kidney and pancreas transplant is the only treatment able to restore euglycemia in patients with type 1 diabetes and selected patients with type 2 diabetes, are now consolidated, rates of transplantation remain low among potential candidates with high levels of preformed anti-HLA antibodies. Most of the data comes from the experience in kidney transplant but can be easily translated to pancreas transplant.

Approximately 30% of patients on the transplant waiting list have evidence of sensitization in the form of alloantibodies, generated from exposure to previous transplants, blood transfusions, pregnancy, or other events. The presence of a panel-reactive antibody level of at least 80% (i.e. a high level of sensitization) creates difficulty in finding matched kidneys from compatible donors, leading to lower rates of transplantation in highly sensitized candidates compared to non-sensitized; the longer waiting times translates in an increased mortality rate. Despite the development of desensitization strategies and the advancement in immunosuppression protocols, it is apparent that transplanting these patients carries an increased risk of acute antibody mediated rejection; 25%-50% of transplants will have an early acute antibody mediated rejection . Most of these rejections can be successfully treated, but a high rate of transplant glomerulopathy and chronic antibody mediated rejection (AMR) leading to accelerated allograft failure is common.

This protocol has been designed to demonstrate the feasibility and efficacy of spleen transplant as a desensitization strategy for highly sensitized patients, potential candidates of kidney or simultaneous kidney pancreas transplant with (positive cross-match by flow cytometry (T or B) or B positive standard cross-match). After obtaining surgical and research consent at a pre-transplant clinic visit, patients will be receiving spleen transplant followed by spleen removal and kidney or simultaneous kidney pancreas transplant. Duration of the subject participation will begin upon consent and will last for one year after the surgery.

Incidence of treated acute rejection (humoral or cellulo-mediated) within the first year (defined as biopsy proven or clinically indicated) will be determined. Graft and patient survival will be monitored and compared with a cohort of highly sensitized patients with similar immunological characteristics, treated with our standard protocol. DSA levels and post-transplant cross-match will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must give written informed consent, and
* Subject is ≥ 18 years of age, and
* Subject is eligible for a kidney or simulateous kidney pancreas transplant, and
* Subjects are highly sensitized (cPRA 98-100%), and
* Subjects have a positive T flow crossmatch

Exclusion Criteria:

* Severe cardiac disease not amenable to intervention
* Clinical significant systemic infection within 30 days prior to transplant
* Life expectancy < 1 Year
* Positive pregnancy test performed < 1 week prior to enrollment or intention to plan a pregnancy in the following year
* Current drug or alcohol abuse
* Uncontrolled, severe psychiatric illness
* Combined transplantation of kidney and other organs

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Rate of successful spleen transplantations/removals that can overcome the immunological barrier of positive T flow crossmatch and allow better results in kidney transplant recipients with high cPRA compared to the standard treatment. | 3 years
  Rate of successful spleen transplantations/removals that can overcome the immunological barrier of positive T flow crossmatch and allow better results in kidney transplant recipients with high cPRA compared to the standard treatment.
Rate of graft success | 3 years
  Rate of graft will be monitored and compared with a cohort of highly sensitized patient and positive T flow crossmatch, treated with our standard protocol.
Rate of patient survival | 3 years
  Rate of patient survival will be monitored and compared with a cohort of highly sensitized patient and positive T flow crossmatch, treated with our standard protocol.

SECONDARY OUTCOMES:
Rate of T flow crossmatch that becomes negative | 3 years
  Rate of T flow crossmatch that becomes negative, leading to less rejections and consequent improved kidney function.

CONTACTS AND LOCATIONS:
Overall Officials: Ivo Tzvetanov, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
No sharing of IPD will be included at this time. We do plan to report our final results after deidentification.